CLINICAL TRIAL: NCT01010204
Title: Varenicline Treatment for Smoking Cessation in Patients With Bipolar Disorder
Acronym: BEST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: K.N. Roy Chengappa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, K.N. Roy Chengappa, Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21MH087928 (NIH); R21MH087928 (NIH)
Record Dates: First submitted 2009-11-05; First posted 2009-11-09 (Estimated); Results first posted 2015-03-12 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2015-04

CONDITIONS: Smoking Cessation; Bipolar Disorder
Keywords: Varenicline; Chantix; Smoking; Bipolar Disorder
MeSH Terms: conditions — Smoking Cessation; Bipolar Disorder; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental): We will be comparing Varenicline to placebo in a double-blind placebo controlled, randomized study.
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): We will be using placebo in a randomized, controlled, and blinded trial to compare to varenicline in subjects with bipolar disorder.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Patients will be randomly assigned to receive either varenicline or placebo for 12 weeks. Patients assigned to varenicline will receive 0.5mg by the oral route once a day for 3 days, followed by 0.5mg twice a day for 4 days. After the first week the dose will be increased to 1mg twice daily for the remainder of the active treatment period of the study, i.e. 11 weeks. Patients assigned to placebo will receive identical looking capsules in a dosage schedule similar to varenicline. Patients will be instructed to take study medication after meals with a glass of water.
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — Patients will be randomly assigned to receive either varenicline or placebo for 12 weeks. Patients assigned to varenicline will receive 0.5mg by the oral route once a day for 3 days, followed by 0.5mg twice a day for 4 days. After the first week the dose will be increased to 1mg twice daily for the remainder of the active treatment period of the study, i.e. 11 weeks. Patients assigned to placebo will receive identical looking capsules in a dosage schedule similar to varenicline. Patients will be instructed to take study medication after meals with a glass of water.
  Other Names: Comparator
  Arms: Placebo

SUMMARY:
The investigators' hypothesis is that add-on varenicline will be effective (versus placebo) in initiating abstinence from smoking in subjects with stable, euthymic bipolar disorder who are motivated to quit smoking within four weeks. This primary outcome will be assessed from randomization to 12 weeks or end of the treatment phase of the study. Secondarily, the investigators also hypothesize that varenicline will prevent relapse in the subsequent 12-weeks follow-up non-treatment phase. Furthermore, the investigators plan to test the effectiveness of varenicline in reducing nicotine withdrawal symptoms or urges to smoke, as well as its safety for use in stable bipolar patients when used as an add-on treatment for smoking cessation.

The investigators plan to test these hypotheses by conducting a randomized, placebo-controlled add-on treatment trial of Chantix with 60 recruited subjects diagnosed with DSM-IV bipolar disorder for a period of three months. The investigators will follow-up with them three months later to evaluate extended abstinence.

DETAILED DESCRIPTION:
OBJECTIVE:

Our primary objective is to determine if adjunctive varenicline will be efficacious (vs. placebo) in initiating abstinence from smoking cigarettes in subjects with stable bipolar disorder who are motivated to quit smoking during a 12-week treatment phase. A secondary outcome is to determine whether those who initiated abstinence during the 12-week treatment phase will maintain abstinence in the subsequent three-month follow-up period off study medications.

Additional outcomes: we plan to test the effectiveness of varenicline in reducing nicotine withdrawal symptoms or urges to smoke, as well as its safety for use in stable bipolar patients when used as an adjunctive treatment for smoking cessation.

RESEARCH PLAN:

We plan to test these hypotheses by conducting a randomized, placebo-controlled, treatment trial of Chantix. Measures of CO levels in expired air (10 ppm or lower), self-reported abstinence, and psychopathology ratings will be used to evaluate primary and secondary outcomes along with safety assessments. Smoking abstinence is defined as 7-day point prevalence of self-reported no smoking verified objectively by expired CO levels of 10 ppm or less, and will be assessed at 12-weeks (or end of treatment phase) as the primary outcome. The same criterion will be used to assess maintenance of abstinence in the non-treatment phase, i.e. at 24 weeks or end of study.

METHODS:

Seventy-six subjects with DSM-IV bipolar disorder will be recruited from Western Psychiatric Institute and Clinic and Dubois Regional Medical Center. Using a 1:1 Randomization, which also takes into account gender, subjects who sign an informed consent document will be randomized to receive Chantix or placebo.

It is expected that 16 of the 76 may not meet inclusion/exclusion criteria, leaving 60 consenting adults aged 18-65 years with DSM-IV bipolar disorder, which will be confirmed by the MINI (Sheehan et al.) Subjects must meet smoking inclusion criteria of smoking 10 or more cigarettes per day. Motivation to quit smoking (score of at least 7 on the Contemplation Ladder Scale) as well as stable mood status (Young Mania Rating Scale score of eight or less, Montgomery Asberg Depression Rating Scale Score of eight or less, with low scores on suicide aggression and psychotic items over a four-week period required. Subjects who have received pharmacological agents for smoking cessation such as bupropion, nicotine replacement treatment, or who have participated in behavioral treatment for smoking cessation more than three months before beginning the study will be permitted to enroll in the study. Anyone experiencing serious side-effects from varenicline in the past or who has already participated in a smoking cessation study with varenicline will be excluded.

Chantix or placebo will be administered using random assignment at a dose of 0.5 mg by mouth for three days, followed by 0.5 mg twice per day for four days. After the first week, the dose will be increased to 1 mg twice daily for 11 weeks. Subjects must be able to tolerate a minimum of 1 mg per day to continue in the study.

Subjects will pick a target date between visit 3 (to permit titration to the target dose of 2 mg per day) and visit 4 to quit smoking. There needs to be at least 24 hours (preferably 48) between the time of the last cigarette usage and visit 4, where a CO measurement will be taken.

Those who are unable to quit at this time will be given an opportunity to pick additional quit dates. All visits will be scheduled a week apart and subjects will continue to take their double-blind medication and receive counseling sessions for smoking cessation. Study medication will be stopped after 12 weeks, and there will be weekly visits to evaluate abstinence.

Some standard psychopathology rating scales and smoking rating scales will be administered to evaluate secondary aims such as the degree of nicotine withdrawal symptoms and the impact of residual symptoms on bipolar disorder. Safety will be assessed through the administration of specific mania and depression rating scales including and the Columbia -Suicide Severity Rating Scale, as well as a comprehensive health assessment. This includes a medical history and evaluation of laboratory measures. Any adverse effects of medication will be assessed by asking questions at each visit and if necessary, contacting the subject by phone outside the scheduled visits.

SIGNIFICANCE The rate of cigarette smoking among people with psychiatric disorders remains exceedingly high; nearly two to four times as high as those in the general population. Patients with bipolar disorder may have the highest rates of smoking as compared with people with other psychiatric diagnoses. To date, there have been no treatment trials of adequate size to measure smoking cessation rates in people with bipolar disorder. If varenicline proves to be an effective in helping people with bipolar disorder to stop smoking, or even to reduce their smoking rates, this could play an important role in improving their health.

ELIGIBILITY:
Subject inclusion criteria

1. DSM IV-TR Bipolar I or II or Bipolar NOS Disorder
2. Ability to provide written informed consent
3. Male or Female patients, all races, ages 18 to 65 years inclusive
4. Negative serum pregnancy test for females of child-bearing potential. Patients must agree to one of the following birth control methods: an oral contraceptive agent, an intrauterine device (IUD), an implantable contraceptive (e.g., Norplant), or an injectable contraceptive (e.g., Depo Provera) for at least 1 month prior to entering the study and will continue its use through at least 30 days after the last dose of study medication or a barrier method of contraception, e.g., condom and/or diaphragm with spermicide while participating in the study through at least 30 days after the last dose of study medication or abstinence.
5. MADRS total scores ≤ 8 (past 4 weeks) (suicidal item, score ≤ 1, past 4 weeks).
6. Y-MRS scores ≤ 8 (past 4 weeks) irritability, speech content, disruptive, or aggressive behavior items score ≤ 3, past 4 weeks)
7. Stable doses of primary bipolar maintenance medication for at least 8 weeks prior to randomization
8. No psychiatric hospitalization or Emergency Room Visits for psychiatric issues in the 6-month period prior to randomization
9. No suicidal attempts or behavior history past 6 months
10. No aggressive or violent acts or behavior by history past 6 months

Subject exclusion criteria

1. Uncontrolled seizure disorders and other neurological disorders including Huntington's Chorea, Multiple Sclerosis, Cerebral Palsy, and stroke (cerebrovascular accident, CVA).
2. Current alcohol or other substance abuse or dependence within the last 3 months (caffeine will be permitted, nicotine dependence is part of inclusion criteria), including a case-by-case evaluation of those who meet remission criteria and who are on long-term substance abuse and/or alcohol abuse treatment.
3. Female patients who are pregnant, lactating or likely to become pregnant in next 6 months
4. Uncontrolled diabetes mellitus, asthma, seizure disorder, uncontrolled hypertension, (uncontrolled hypertension is defined as Systolic BP > 150 mm or Hg or diastolic BP > 95 mm or Hg on 2 consecutive BP readings 15 minutes apart at the time of screening) or unstable medical illness. Moderate to severe renal disease - moderate renal failure is defined as serum Creatinine >1.3 mg/dl in women and > 1.5 mg/dl in men, at the time of screening.
5. Severe dizziness or fainting due to orthostatic blood pressure changes
6. Known hypersensitivity to varenicline
7. Current use of cimetidine
8. Current treatment with heparin, warfarin, or lidocaine
9. Comorbid psychiatric condition diagnosed within the last three months.

Subject smoking inclusion criteria

1. Score of 7 or greater on the Contemplation Ladder, and willing to pick a target quit date within the next 4 weeks.
2. Smoke > 10 cigarettes per day.
3. Expired breath CO level > 10 ppm at screening and randomization.
4. No use of smoking cessation medication and/or behavioral treatment for smoking cessation in the past three months.
5. No current use of any nicotine replacement treatment.
6. Not using any tobacco products other than cigarettes.
7. No current treatment for smoking cessation (hypnosis, acupuncture, others).
8. No current use or past treatment failure with varenicline.
9. No current treatment with bupropion for smoking cessation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K.N. Roy Chengappa, Principal Investigator — University of Pittsburgh School of Medicine Department of Psychiatry
Locations (2):
- United States (2):
  - Dubois Regional Medical Center, DuBois, Pennsylvania
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Chengappa KN, Perkins KA, Brar JS, Schlicht PJ, Turkin SR, Hetrick ML, Levine MD, George TP. Varenicline for smoking cessation in bipolar disorder: a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2014 Jul;75(7):765-72. doi: 10.4088/JCP.13m08756. PMID 25006684
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: We will be comparing Varenicline to placebo in a double-blind placebo controlled, randomized study.
  Varenicline (Chantix): Patients will be randomly assigned to receive either varenicline or placebo for 12 weeks. Patients assigned to varenicline will receive 0.5mg by the oral route once a day for 3 days, followed by 0.5mg twice a day for 4 days. After the first week the dose will be increased to 1mg twice daily for the remainder of the active treatment period of the study, i.e. 11 weeks. Patients assigned to placebo will receive identical looking capsules in a dosage schedule similar to varenicline. Patients will be instructed to take study medication after meals with a glass of water.
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 31 | 29
Completed | 24 | 20
Not Completed | 7 | 9
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — psychiatric hospitalization | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (10.3) | 46.2 (8.5) | 45.95 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 20 | 21 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 7-day Prevalence of Abstinence From Cigarette Smoking at 12 Weeks
Description: To evaluate the efficacy of varenicline treatment added to standard behavioral treatment for smoking abstinence at 12 weeks
Time Frame: 12 weeks
Population: bipolar subjects
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 31 | 29
participants | 15 | 3

2. Primary Outcome: 7 Day Prevalence of Abstinence From Cigarette Smoking at 24 Weeks
Description: To evaluate the efficacy of varenicline treatment added to standard behavioral treatment for smoking abstinence
Time Frame: 24 weeks
Population: bipolar patients
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 31 | 29
participants | 6 | 2

3. Secondary Outcome: Participants Experiencing Neuropsychiatric Events
Description: Evaluate the safety of varenicline in treatment-emergent hypomania, mania, mixed or depressed episodes or being associated suicidal or aggressive behavior or psychotic symptoms when used as adjunctive treatment in participants with bipolar disorder.
Time Frame: 24 weeks
Population: Bipolar Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 31 | 29
Participants | 7 | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 6/31 | 4/29
Other Adverse Events (participants affected / at risk) | 29/31 | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=31) | Placebo (N=29)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
exacerbation of anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
agitation, hostility, alcohol drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
asthma with acute exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
alcohol intoxication (Psychiatric disorders) | 0 (0) | 1 (1)
upper left arm weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
chest pain, left hand numbness (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=31) | Placebo (N=29)
diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
constipation (Gastrointestinal disorders) | 7 (7) | 5 (5)
dry mouth (General disorders) | 9 (9) | 9 (9)
flatulance (Gastrointestinal disorders) | 11 (11) | 11 (11)
vomiting (Gastrointestinal disorders) | 3 (3) | 6 (6)
nausea (Gastrointestinal disorders) | 13 (13) | 9 (9)
heart burn (Gastrointestinal disorders) | 7 (7) | 6 (6)
abdominal pain (Gastrointestinal disorders) | 6 (6) | 6 (6)
gastroesophageal reflux (Gastrointestinal disorders) | 7 (7) | 2 (2)
depressed mood (Psychiatric disorders) | 8 (8) | 2 (2)
anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
mood swings (Psychiatric disorders) | 2 (2) | 1 (1)
insomnia (Psychiatric disorders) | 14 (14) | 8 (8)
abnormal dreams (Psychiatric disorders) | 18 (18) | 9 (9)
suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
somnolence (Nervous system disorders) | 2 (2) | 1 (1)
headache (Nervous system disorders) | 11 (11) | 12 (12)
dizziness (Nervous system disorders) | 2 (2) | 1 (1)
bad taste (Nervous system disorders) | 4 (4) | 2 (2)
arthralgia/pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
fatigue/lethargy (General disorders) | 8 (8) | 5 (5)
asthenia-weakness (General disorders) | 1 (1) | 4 (4)
runny nose (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
increased appetite (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 6 (6)
weight gain (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
weight loss (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No